CLINICAL TRIAL: NCT02287246
Title: Efficacy of Extended-Release Liposomal Bupivacaine for Post-Operative Pain Management Following Urogynecologic Surgery: A Prospective, Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Efficacy of Extended-Release Liposomal Bupivacaine for Post-Operative Urogynecologic Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christy Jones, Principal Investigator, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 399635
Record Dates: First submitted 2014-11-05; First posted 2014-11-10 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extended-Release liposomal bupivacaine (Experimental): 20mL Extended-release liposomal bupivacaine injected into the posterior vaginal wall following surgery
  Interventions: Drug: Extended-Release liposomal bupivacaine (Exparel)
- Placebo (normal saline) (Active Comparator): 20mL normal saline injected into the posterior vaginal wall following surgery
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Extended-Release liposomal bupivacaine (Exparel) — 20mL
  Other Names: Exparel
  Arms: Extended-Release liposomal bupivacaine
Drug: Normal saline — 20mL
  Arms: Placebo (normal saline)

SUMMARY:
To study post-operative efficacy of Exparel® for pain control in patients undergoing any Urogynecology surgery involving the posterior vaginal wall using a randomized, double-blinded placebo controlled trial.

DETAILED DESCRIPTION:
Effective post-operative pain management is a crucial component of a patient's surgical course following Urogynecologic surgery. Narcotics are the cornerstone for post-operative analgesia with a frequent re-dosing requirement, a lengthy list of side effects and adverse reaction risks5. The colorectal, orthopedic and general surgery literatures have reported on an extended-release bupivacaine liposomal injection, Exparel®, which remarkably reduces acute post-operative pain; however, this medication has not yet been reported within Urogynecology literature.

We propose a prospective, randomized, double blind, placebo controlled trial with 120 subjects recruited from the WRNMMC Urogynecology Clinic to study post-operative efficacy of Exparel® for pain control in patients undergoing Urogynecology surgery involving the posterior vaginal wall. Subjects will be randomized to receive either 20mL of extended-release bupivacaine or 20mL placebo.

The primary objective of the trial will be to evaluate the cumulative post-operative vaginal pain using front side of Defense and Veterans Pain Rating Scale16 at days 1 and 3 post-procedure.. We hypothesize a 30% difference in post-operative pain measurements between the active medication group and placebo group.

Additional objectives of this study are to evaluate vaginal pain on post-operative day 7, total medication usage on days 1, 3 and 7 and any post-operative voiding dysfunction, comparing the study group to the control.

ELIGIBILITY:
Inclusion Criteria:

Females >18 years of age undergoing Urogynecologic surgery involving the posterior vaginal wall mucosa or muscularis (including but not limited to posterior colporrhaphy, colpocleisis, sphincter repair, sphincteroplasty, perineoplasty) at Walter Reed National Military Medical Center. Patients must be able to read and understand written English or have an appropriate certified medical translator available.

Exclusion Criteria:

Known allergy to amide local anesthetics Unstable cardiac arrhythmia Hepatic impairment (including but not limited to patients under the care of their physician for severe hepatic disease, cirrhosis or hepatic cancer) Known pregnancy at time of surgery (pregnancy test morning of surgery if applicable) Regular use of narcotic pain medication, defined as use on most days of week at any time in the three months prior to surgery Significant history of opioid or alcohol abuse or addiction (requiring treatment) Concurrent pain management requiring the use of epidural anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Cumulative post-operative pain control | Post operative day 1 and 3
  The primary objective of the trial will be to evaluate the cumulative post-operative vaginal pain using front side of Defense and Veterans Pain Rating Scale16 at days 1 and 3 post-procedure.. We hypothesize a 30% difference in post-operative pain measurements between the active medication group and placebo group.

SECONDARY OUTCOMES:
Evaluate vaginal pain on Post-operative day 7 | Post-operative day 7
  Additional objectives of this study are to evaluate vaginal pain on post-operative day 7, total medication usage on days 1, 3 and 7 and any post-operative voiding dysfunction, comparing the study group to the control.

CONTACTS AND LOCATIONS:
Overall Officials: Christin L Jones, DO, Principal Investigator — WRNMMC
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Planning to publish once completed